CLINICAL TRIAL: NCT00002423
Title: A Phase II, Open-Label Trial for Treatment of HIV Infection in Subjects Who Have Failed Initial Combination Therapy With Regimens Containing Indinavir or Nelfinavir: Combination Therapy With 3TC (150 Mg BID), Abacavir (300 Mg BID) and Amprenavir (1200 Mg BID) Plus Either Nelfinavir (1250 Mg BID) or Indinavir (800 Mg TID) for 48 Weeks
Brief Title: A Study to Compare Two Anti-HIV Drug Combinations That Include Amprenavir in HIV-Infected Patients Who Have Failed Anti-HIV Drug Combinations That Did Not Include Amprenavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 264M; PRO20005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Lamivudine; Indinavir; Nelfinavir; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; amprenavir; Nelfinavir; Lamivudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Lamivudine

SUMMARY:
This study will compare the safety and effectiveness of two anti-HIV drug combinations in fighting HIV infection in patients whose viral loads (levels of HIV in the blood) rose with other anti-HIV drug treatments.

DETAILED DESCRIPTION:
Patients experiencing virologic failure while receiving an IDV-containing antiretroviral regimen will receive the 3TC/ABC/APV/NFV combination. Patients experiencing virologic failure while receiving an NFV-containing antiretroviral regimen will receive the 3TC/ABC/APV/IDV combination.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this trial if you:

* Are HIV-positive.
* Are 13 years of age or older.
* Are currently taking anti-HIV drugs, 1 of which must be NFV or IDV, and have taken these same drugs for at least 12 weeks.
* In the last 16 weeks your viral load (level of HIV in the blood) dropped below 400 copies/ml and has since increased to at least 1,000 copies/ml, even though you continue to take your anti-HIV drugs.
* Have the written consent of a parent or legal guardian if you are under age 18.
* Agree to practice abstinence or use effective barrier methods of birth control (unless you are physically incapable of becoming pregnant).
* Are willing to complete the 48-week study.

Exclusion Criteria

You will not be eligible for this trial if you:

* Have ever taken the following anti-HIV drugs: ABC, APV, efavirenz (EFV), delavirdine (DLV), nevirapine (NVP), or loviride.
* Have certain AIDS-related infections or diseases, have other serious medical conditions such as diabetes and certain types of heart trouble, or have a history of lymphoma.
* Have had certain types of hepatitis in the past 6 months.
* Have received an HIV vaccine in the past 3 months or a flu vaccine in the past 30 days.
* Have certain digestion problems that make it difficult to take anti-HIV drugs by mouth.
* Have received certain other drugs or treatments in the past 30 days, or will need certain drugs or treatments during the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Saint Francis Mem Hosp, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Natl Institute of Allergy and Infectious Diseases, Bethesda, Maryland
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Bentley-Salick Med Practice, New York, New York
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon